CLINICAL TRIAL: NCT06542926
Title: Electronic Dataset of NON-COlorectal Liver METastases Undergoing Liver Resection
Brief Title: NON-COlorectal Liver METastases Undergoing Liver Resection
Acronym: NONCOLMET
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Matteo Donadon, Professor of Surgery, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: NONCOLMET01
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Liver Metastases
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: liver resection — Resection of non-colorectal liver metastases
  Other Names: hepatectomy

SUMMARY:
Liver metastases (LM) are common in various types of malignant diseases, either at the diagnosis of the primary tumour or at a later time point. While the resection of colorectal LM (CRLM) is a well-established procedure, with survival rates superior to chemotherapy alone, controversial data still exist on liver resection for non-colorectal LM (NCRLM) (2, 3). These patients comprise a diverse and heterogeneous group usually excluded from surgery due to advanced tumour stage or the presence of concomitant extrahepatic disease. To date, no randomized clinical trial on the surgical treatment of NCRLM has been conducted, and only few retrospective reports are available.The scope of this research project is to develop a large registry of patients undergoing liver surgery for non-colorectal liver metastases.

ELIGIBILITY:
Inclusion criteria:

* Signature informed consent
* Age ≥ 18 years
* Histologically confirmed diagnosis of NCRLM (first diagnosis or relapse)
* Liver resection performed.

Exclusion criteria

* ASA IV
* Severe psychiatric pathology
* Unable to follow a clinical examination pattern during observation.
* Patient submitted exclusively to interventional locoregional procedures other than liver resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis, based on imaging methods and histologically confirmed, of NCRLM, consecutively referred to centres with expertise in hepatobiliary surgery will be evaluated for inclusion. For the diagnosis and staging of disease the participating centres will refer to the guidelines for NCRLM, together with the established clinical habits present in each centre
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From date of enrollment until the date of death from any cause assessed up to 36 months
  Overall Survival defined as the time elapsed between the date of resective surgery and the date of death for any reason. Patients who are surviving at the end of observation will be considered "censored" at the date of the last available follow-up.

SECONDARY OUTCOMES:
Disease-free Survival | From date of enrollement until the date of first documented progression assessed up to 36 months
  Disease-free Survival defined as the time from resective surgery to the date of first relapse or last available follow-up, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Donadon, MD, PhD, Principal Investigator — AOU della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: No